CLINICAL TRIAL: NCT00966043
Title: Prevalence of Genetic Polymorphisms in Genes Coding for Tamoxifen Metabolising Enzymes, in Postmenopausal ER-positive Breast Cancer Patients According to Uterine and Biochemical Changes and Tolerability of Tamoxifen.
Brief Title: Prevalence of Genetic Polymorphisms in Genes Coding for Tamoxifen Metabolising Enzymes
Acronym: CYPTAMBRUT-3
Status: Completed | Type: Observational
Sponsor: Vlaamse Vereniging voor Obstetrie en Gynaecologie (Other)
Responsible Party: Sponsor
Other Study IDs: Eudract 2009-010059-28.; S 51521
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
CYPTAM-BRUT 3 is a prospective, multicentric study in Belgium within the CYPTAM study of the Leiden University Medical Center (NTR1509) including postmenopausal women receiving tamoxifen for estrogen-receptor positive breast cancer in the adjuvant setting. The primary endpoint is the difference in uterine changes between women with a normal versus low TAS after 3 months of tamoxifen use. Secondary endpoints are serum metabolite concentrations, serum follicle-stimulating hormone level, serum sex hormone-binding globulin level and menopausal symptoms. These patients are registered in the Leiden protocol with time to breast cancer event as primary endpoint.

DETAILED DESCRIPTION:
We will study the impact of the 'tamoxifen activity score' - based on functional genetic polymorphisms for tamoxifen metabolism and the use of drugs that interfere with tamoxifen-against tamoxifen related endpoints like uterine changes and subjective menopausal symptoms.

The prevalence of genetic polymorphisms in the CYP2D6 and other genes and differences in usage of drugs interacting with tamoxifen metabolism will be compared between women with and those without endometrial thickening on one hand and between women with and those without hot flashes on the other hand. Tamoxifen use in adjuvant setting.

* "Tamoxifen activity score" (23): The endpoints will be correlated with a predefined 'tamoxifen activity score' which is based on the presence of single nucleotide polymorphisms (SNP) in relevant genes combined with the effect of well known drugs that interfere with the metabolism of tamoxifen. The 'tamoxifen activity score' has been associated with tamoxifen compliance by a group in the US (23). The score will be adapted to the Belgian situation based on the prevalence of these SNPs in a Belgian population of volunteers for blood donation and consecutive breast cancer patients.
* The study setting are postmenopausal women with an early ER- positive breast cancer and not previously treated with an endocrine agent or hormone replacement therapy, with an intact uterus and clearly measurable thin endometrium/uterus. N =250

ELIGIBILITY:
Inclusion Criteria:

* Female > 18 years of age
* Written and voluntary informed consent understood signed and dated
* Histologically or cytologically confirmed measurable invasive adenocarcinoma of the breast, amenable to curative therapy.
* Patients must be postmenopausal as defined by criteria in appendix 1.
* Breast cancer should be considered as oestrogen receptor positive by the clinician using immunohistochemistry readings as is standard procedure for local pathologist
* Prior endocrine tamoxifen therapy is not allowed
* Patients are not previously treated with an endocrine agent or hormone replacement therapy needs being stopped for at least 6 months.
* Prior chemotherapy and radiotherapy is allowed
* Adequate renal and liver function Serum creatinine and serum bilirubin ≤ 1.5 X ULN Serum ALT and AST ≤ 2.5 X ULN (or ≤ 5 in case of liver metastases)
* Serum calcium should be ≤ 11,6 mg/dl
* ECOG performance status 0,1,2 (appendix 2)

Exclusion Criteria:

* Male
* Life threatening disease requiring a quick response (eg, extensive hepatic or pulmonary involvement)
* Use of any endocrine treatment or recent/current use of hormone replacement therapy.
* Contra indication for tamoxifen: history of DVT/vaginal bleeding of unknown origin
* Dementia
* History of other malignancy that may interfere with at least 6 months of tamoxifen therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal female breast cancer patients starting adjuvant tamoxifen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
change in endometrial thickness or uterine volume | 3-6 months

SECONDARY OUTCOMES:
Tolerability of tamoxifen-HRQoL questionnaire | 3-6 months
Vaginal bleeding | 3-6 months
Biochemical changes | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Neven, Principal Investigator — UZ Leuven
Locations (11):
- Belgium (11):
  - AZ St-Maarten, Duffel, Antwerpen
  - AZ St-Nikolaas, St-Niklaas, Antwerpen
  - Ziekenhuizen Oost-Limburg Camus St-Jan, Genk, Limburg
  - AZ St-Blasius, Dendermonde, Ookst-Vlaanderen
  - Maria-Middelares, Ghent, Oost-Vlaanderen
  - UZ, Ghent, Oost-Vlaanderen
  - UZ, Leuven, Vlaams-Brabant
  - Heilig-Hart Ziekenhuis, Roeselare, West-Vlaanderen
  - Institut Bordet, Brussels
  - UZ, Brussels
  - UCL, Brussels